CLINICAL TRIAL: NCT02695381
Title: A Randomized, Double-blind, Multiple-dose, Placebo-controlled Study to Evaluate the Efficacy and Safety of Etodolac-lidocaine Patch Applied Once Daily in Subjects Experiencing Acute Delayed Onset Muscle Soreness
Brief Title: Etodolac-lidocaine Patch in Subjects Experiencing Acute Delayed Onset Muscle Soreness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDRx USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MRX-7EAT-1010
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Acute Delayed Onset Muscle Soreness (DOMS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etodolac-lidocaine Topical Patch (Experimental): Therapy with experimental drug
  Interventions: Drug: Etodolac-lidocaine topical patch
- Placebo (Placebo Comparator): Therapy with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etodolac-lidocaine topical patch — Once daily
  Other Names: Etoreat
  Arms: Etodolac-lidocaine Topical Patch
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
This study evaluate the efficacy and safety of Etodolac-lidocaine topical patch applied one time daily when compared with placebo in the treatment of acute Delayed Onset Muscle Soreness (DOMS) of the upper limbs.

ELIGIBILITY:
Inclusion Criteria:

* Have not engaged in significant upper extremity fitness activities for more than two times per week for ≥ 2 consecutive weeks in the past 6 months prior to screening.
* Subject has a body mass index of between 18 and 30 kg/m2, inclusive.
* Subjects who report a pain with movement score in both arms of at least 5 (based on a 0-10 NRS) secondary to DOMS approximately 24 to 30 hours after each arm was exercised.

Exclusion Criteria:

* Presence of another painful physical condition that, in the opinion of the Investigator, may confound study assessments.
* Use of pain medication (including anti-inflammatory drugs) prior to the Exercise Visit until 72 hours after randomization.
* Use of any corticosteroids (oral, injectable, topical, inhaled) from before the Exercise Visit until randomization. Corticosteroids must be washed out by at least 3 days before the Exercise Visit.
* Chronic or acute renal or hepatic disorder, inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) or a significant coagulation defect.
* History of allergy (cutaneous or systemic), asthma, hypersensitivity to any of the following: etodolac, lidocaine, paracetamol (acetaminophen), acetylsalicylic acid, salicylic acid, other NSAID, other local anesthetic, known intolerance (cutaneous or systemic) to any of the ingredients in the patch.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Sum of the time-weighted differences from baseline in pain intensity with movement (SPIDMove) over 0-24 hours post-T0 (SPIDMove 0-24 hours). | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paulette Saddler, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No